CLINICAL TRIAL: NCT01036438
Title: A Double-blind, Comparative, Superiority, Multi-centre Investigation Evaluating the Efficacy of an Absorbent Foam Dressing Containing Silver (Mepilex Ag) Versus the Same Dressing Without Silver Used on Subjects With Venous Leg Ulcers or Mixed Ulcers
Brief Title: Evaluating the Efficacy of an Absorbent Foam Dressing Containing Silver (Mepilex Ag) Versus the Same Dressing Without Silver Used on Subjects With Venous Leg Ulcers or Mixed Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUMA 416
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2013-12

CONDITIONS: Venous Leg Ulcers; Mixed Leg Ulcers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepilex product (Placebo Comparator)
  Interventions: Device: Mepilex without Ag
- Mepilex Ag (Active Comparator)
  Interventions: Device: Mepilex Ag

INTERVENTIONS:
Device: Mepilex Ag — Mepilex is designed for a wide range of exuding wounds such as leg and foot ulcers, pressure ulcers and traumatic wounds, e.g. skin tears and secondary healing wounds.
  Arms: Mepilex Ag
Device: Mepilex without Ag — Mepilex is designed for a wide range of exuding wounds such as leg and foot ulcers, pressure ulcers and traumatic wounds, e.g. skin tears and secondary healing wounds.
  Arms: Mepilex product

SUMMARY:
Compare the efficacy of using an absorbent foam silver dressing (Mepilex Ag) versus the equivalent dressing without silver in subjects suffering from venous leg ulcer or mixed ulcer with an ABPI ≥ 0.8 and with inflammatory signs. Efficacy will be defined as absolute wound size reduction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with colonised/ local infection in a venous leg ulcer or mixed leg ulcer with an ABPI ≥ 0,8 and < 1.3
* A history of an appropriate compression therapy for at least 2 weeks prior to randomisation
* Subjects with colonised/local infection presenting with three of five following specified signs:

  * pain between dressing changes
  * exuding wounds
  * erythema on peri-wound skin
  * oedema
  * odour
* An ulcer size of at least 4 cm2 and a maximum size witch could be covered by one investigational product of 15x15 cm.
* Ulcer duration 6 weeks to 1 year
* In case of multiple ulcers: target ulcer must be at least 3 cm distant from other ulcers.
* Both gender with an age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* > 10% necrotic (black) or fibrinous (yellow) tissue covering the wound bed
* Infected wounds in need of systemic antibiotic treatment
* Use of anti-microbial dressings or topical agents such as antiseptics, local antibiotics and steroids within 7 days from inclusion on the wound intended to be included
* Previous treatment with silver product 2 weeks prior to inclusion
* Previous treatment with MepilexAg® on the target ulcer
* Use of systemic antibiotics for any reason during the previous 7 days
* Venous surgery 2 weeks prior to inclusion or planned surgery within 8 weeks after inclusion
* Diagnosed underlying disease(s) (e.g. HIV/AIDS, cancer/malignancy and severe anaemia) judged by the investigator to be a potential interference in the wound evaluation
* Subjects with poorly controlled diabetes mellitus i.e. HbA1c >8%
* Subjects treated with systemic immunosuppressive or glucocorticosteroids, except subjects taking occasional doses or doses less than 10mg prednisolon/day or equivalent. Subjects inhaling glucocorticosteroids for asthma should not be excluded.
* Known allergy/hypersensitivity to any of the components of the investigation products.
* Subjects with physical and/or mental conditions that are not expected to comply with the investigation due to poor medical condition
* Participation in other clinical investigation(s) within 1 month prior to start of the investigation.
* Previously randomised to this investigation.
* Life expectance of the subject less than 3 months
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2009-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Meaume, Dr, Principal Investigator — Hopital Rotchild - Jean Rostand, Paris
Locations (44):
- Czechia (11):
  - Nemocnice Jihlava, Jihlava, Jihlava
  - Krajská nemocnice Liberec, Liberec, Liberec
  - chirugické oddělení, Fakultní nemocnice Královské Vinohrady, Prague, Prague
  - Nemocnice Podlesí a.s., Třinec, Třinec
  - Uherskohradišťská nemocnice a. s., Uherské Hradiště, Uherské Hradiště
  - Fakultní nemocnice U svate Anny, St. Anne´s University Hospital, Brno
  - Dermatovenerologická klinika, University Hospital Bohunice,, Brno
  - Dermatovenerologická klinike, Univerzita Karlova, Pilsen
  - Fakultní nemocnice Na Bulovce, Prague
  - Masarykova Hospital, Dermatology dept., Ústí nad Labem
  - Dermatovenerologie Rendlová s.r.o., České Budějovice, České Budějovice
- France (23):
  - Polyclinique de Picardie Service d'Angiologie Phlébologie, Amiens, Amiens
  - Hôpital privé d'Antony Service de Dermatologie, Antony, Antony
  - Hôpital Saint Jacques - CHU Besançon, Besançon, Besançon
  - Résidence le Bristol, Boulogne-sur-Mer, Boulogne-sur-mer
  - CHU Le Bocage Service Dermatologie, Dijon, Dijon Cedex
  - Hôpital Albert Michallon Service de médecine vasculaire, Grenoble, Grenoble Cedex 9
  - CHG La Roche-sur-Yon Service de D'Angiologie,Les Oudairies, La Roche-sur-Yon, La Roche-sur-Yon
  - Centre Hospitalier le Mans Service de Dermatologie, Le Mans, Le Mans Cedex 9
  - Pharmacie Centrale-Service Arsenal, Nantes, Nantes
  - APHP Hôpital Lariboisère, Paris, Paris
  - Hôpital Saint Joseph, Paris, Paris
  - Cabinet d'Angiologie, 1 bis rue de Salgareda, Saint-Alban, Saint Alban
  - Dermatology Department, University Hospital, Hopital Sud, Amiens
  - Service de Dermatologie, Centre Hospitalier Regional Universitaire, Caen
  - Cabinet D'Angeiologie, Lille
  - Hopital Maringer-Villemin- Fournier, Nancy
  - Hôpital Rotchild - Jean Rostand, Paris
  - Hopital Robert Debré Service de Dermatologie, Reims
  - Hopital Charles Nicolle, Rouen
  - Maison de Santé Protestante de Bordeaux-Bagatelle, Talence
  - Hopital Beauregard / Secrétariat de Dermatologie, Thionville
  - Service de dermatologie, Toulon
  - Clinique Pasteur, Toulouse
- Germany (8):
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck, Germany
  - Universtätsmedizin Charité Klinik für Dermatologie, Allergologie und Venerologie, Berlin
  - Venenzentrum der Dermatologischen und Gefäßchirurgischen Kliniken -, Bochum
  - Universitätsklinikum Hamburg-Eppedorf, Hamburg
  - Bramfelder Chaussee 200, Hamburg
  - Universität klinikum Jena, Klinik für dermatologie und dermatologische, Jena
  - University Hospital Regensburg, Regensburg
  - Universitäts-Hautklinik, Tübingen
- Netherlands (2):
  - Dermatology department, Amsterdam
  - St. Antonius Ziekenhuis, Utrecht

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mepilex Product | Mepilex Ag
Started | 101 | 100
Completed | 91 | 90
Not Completed | 10 | 10
Not completed — Adverse Event | 7 | 8
Not completed — Death | 0 | 1
Not completed — No effect of study treatment | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepilex Product | Mepilex Ag | Total
Number analyzed (Participants) | 101 | 100 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (14.9) | 68.4 (13.4) | 67.5 (14.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 42 | 89
  >=65 years | 54 | 58 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 58 | 112
  Male | 47 | 42 | 89
Region of Enrollment [Number; unit: participants]
  France | 25 | 26 | 51
  Czech Republic | 47 | 47 | 94
  Netherlands | 1 | 1 | 2
  Germany | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Will be Defined as Absolute Wound Size Reduction.
Description: Efficacy will be defined as absolute wound size reduction.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Mepilex Product | Mepilex Ag
Number analyzed (Participants) | 101 | 100
cm2 | -4.65 (15.43) | -5.09 (14.23)

2. Secondary Outcome: Change in Inflammatory Signs
Description: Change in inflammatory signs
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Mepilex Product | Mepilex Ag
Serious Adverse Events (participants affected / at risk) | 2/101 | 4/100
Other Adverse Events (participants affected / at risk) | 28/101 | 20/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Product (N=101) | Mepilex Ag (N=100)
Aggravation of ulcus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Aggravation of ulcus, no antibiotics, mailfunktion of dressing.
Erysephilas needing hospitalisation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Erysephilas needing hospitalisation,
Pain on left arm /shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute exacerbation of psoriasis vulgaris (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac decompensation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mepilex Product (N=101) | Mepilex Ag (N=100)
Adverse event related to the ulcer (Skin and subcutaneous tissue disorders) | 19 | 14
Other Adverse Event not related to the ulcer (Investigations) | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less